CLINICAL TRIAL: NCT01712217
Title: A Study of HSP90 Inhibitor AT13387 Alone and in Combination With Crizotinib in the Treatment of Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of AT13387 in Patients With Non-Small Cell Lung Cancer (NSCLC) Alone and in Combination With Crizotinib
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT13387-05; 2012-001575-37 (EudraCT Number)
Record Dates: First submitted 2012-10-11; First posted 2012-10-23 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Non-small Cell Lung Cancer(NSCLC)
Keywords: Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — (2,4-dihydroxy-5-isopropylphenyl)-(5-(4-methylpiperazin-1-ylmethyl)-1,3-dihydroisoindol-2-yl)methanone; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AT13387 and Crizotinib (Experimental): Part A is a single-arm, Phase 1, open-label, dose-escalation design in patients with NSCLC who have already been receiving crizotinib 250 mg by mouth (PO) twice daily (BID) for at least 8 weeks and are still tolerating treatment at that dose. Patients will continue treatment with crizotinib + escalating doses of AT13387 IV weekly for 3 weeks in a 4-week cycle. Each cohort will consist of at least 6 patients until the maximum tolerated dose (MTD) is reached. An additional 12 patients will be treated at the MTD level of AT13387 in combination with crizotinib to confirm the safety profile of the combination at that dose level.
  Interventions: Drug: AT13387; Drug: Crizotinib
- Crizotinib versus crizotinib + AT13387 (Active Comparator): Part B is a Phase 2, open-label, randomized continuation design comparing crizotinib alone versus the combination of crizotinib + AT13387 at the MTD established in Part A. Part B will enroll 128 patients with NSCLC who have been treated with crizotinib for at least 8 weeks and are still tolerating treatment without evidence of disease progression.
  Interventions: Drug: AT13387; Drug: Crizotinib
- AT13387 or AT13387 + crizotinib (Active Comparator): Part C is an open-label, randomized, Phase 2, Simon's 2-stage design of AT13387 administered alone once weekly for 3 weeks (QW×3) or in combination with crizotinib at the MTD established in Part A.
  Interventions: Drug: AT13387; Drug: Crizotinib

INTERVENTIONS:
Drug: AT13387 — HSP90 inhibitor
Drug: Crizotinib — ALK (anaplastic lymphoma kinase) and ROS1 (c-ros oncogene1, receptor tyrosine kinase) inhibitor
  Other Names: Xalkori

SUMMARY:
The purpose of the study is to evaluate safety and efficacy of AT13387 Alone and in Combination with Crizotinib in the Treatment of Non-small Cell Lung Cancer.

DETAILED DESCRIPTION:
This is a 3-part phase 1-2 study in patients with anaplastic lymphoma kinase (ALK) + or other potentially crizotinib-sensitive NSCLC who have been receiving crizotinib. Part A is a single-arm, Phase 1, open-label, dose escalation design in patients with NSCLC who have already been receiving crizotinib for at least 8 weeks and continue to tolerate therapy. Part B is a Phase 2, open-label, randomized continuation design comparing crizotinib alone versus the combination of crizotinib + AT13387 at the maximum tolerated dose established in Part A. Part C is an open-label, randomized, Phase 2, Simon's 2 stage design evaluating single agent AT13387 or combination AT13387 + crizotinib at the MTD established in Part A in patients who progressed on crizotinib at any time.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18 years of age or older
2. Must have Non-small Cell Lung Cancer with ALK+ mutation or other mutations or rearrangements potentially sensitive to crizotinib
3. Measurable disease
4. Must have been receiving or have received crizotinib
5. Have adequate cardiac, bone marrow, liver and kidney function
6. Must be willing and able to provide written informed consent and comply with the protocol and study procedures

Exclusion Criteria:

1. Prior anti-cancer treatment with any HSP90 inhibitor
2. Have received chemotherapy, radiation therapy or other anticancer treatment other than crizotinib within 3 weeks prior to the first dose of study drug
3. Prior malignancy other than adequately treated basal or squamous cell carcinoma of the skin, superficial bladder cancer, low-grade cervical cancer, non-metastatic prostate cancer, or have been disease-free for at least 3 years
4. Abnormal heart function
5. Presence of a life-threatening illness, medical condition, organ system dysfunction, or other factors
6. Hypersensitivity of AT13387 or other components of the drug product
7. Treatment with an investigational drug within 3 weeks prior to the first dose of study drug
8. Severe systemic diseases or active uncontrolled infections
9. Known history of human immunodeficiency virus (HIV) or seropositive test for hepatitis C virus or hepatitis B virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-10; Primary Completion 2016-12 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Part A: The incidence of dose limiting toxicities when AT13387 is administered in combination with crizotinib. | 12 months
  - Number of patients with adverse events
Part B: The comparison of objective response rate by RECIST 1.1 between crizotinib alone and the combination of crizotinib + AT13387. | 18 months
  - Change in tumor measurements by RECIST 1.1 every 8 weeks
Part C: The objective overall response rate for AT13387 alone and the objective response rate (CR+PR) for AT13387 + crizotinib at Stage 1 and Stage 2 of the Simon's 2-stage design. | 18 months
  - Change in tumor measurements by RECIST 1.1 every 8 weeks

SECONDARY OUTCOMES:
Part A: Pharmacokinetics of combination treatment with AT13387 and crizotinib | 12 months
  * Area under the plasma concentration versus time curve (AUC) of AT13387 and crizotinib alone and in combination Week 4
  * Maximum concentration (Cmax) OF AT13387 and crizotinib alone and in combination by Week 4
Part A: Assess antitumor activity of crizotinib + AT13387 combination, circulating tumor cells (CTCs) response, progression free survival (PFS) and overall survival (OS). | 12 months
  * Change in tumor measurements by RECIST 1.1 every 8 weeks
  * Change in CTCs from baseline every 4 weeks
  * Assessment of PFS and OS as measured by weeks
Part B: Assess safety of AT13387 in combination with crizotinib; compare PFS and OS between crizotinib and crizotinib + AT13387; and assess overall response rate (CR + PR) in crizotinib patients who crossover to crizotinib + AT13387 | 18 months
  * Number of patients with adverse events
  * PFS and OS as measured in weeks
  * Response rate as measured by RECIST 1.1 every 8 weeks
Part C: Assess safety of AT13387 alone and in combination with crizotinib who progressed on crizotinib treatment; and compare the PFS and OS of AT13387 administered alone or in combination with crizotinib | 18 months
  * Number of patients with adverse events
  * PFS and OS as measured in weeks

CONTACTS AND LOCATIONS:
Locations (65):
- United States (38):
  - Mayo Clinic-Scottsdale, Scottsdale, Arizona
  - University of California, San Diego Medical Center, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Sharp Clinical Oncology Research-Sharp Memorial Hospital, San Diego, California
  - Innovative Clinical Research Institute, Whittier, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University School of Medicine-Yale Cancer Center, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Florida Hospital Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Northwestern University The Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University Melvin and and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center Eppley Cancer Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Oncology Hematology in Cincinnati, Cincinnati, Ohio
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - The Pennsylvania State University-Penn State, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The West Clinic, Germantown, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin-Carbone Cancer Center, Madison, Wisconsin
- Canada (5):
  - Atlantic Clinical Cancer Research Unit, Halifax, Nova Scotia
  - McGill University Health Center, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie De Quebec, Sainte-Foy, Quebec
  - Princess Margaret Hospital, Toronto, Ontario
  - Cancer Care Manitoba, Winnipeg
- France (10):
  - Centre Hospitalier Regional Universitaire Besancon, Besançon
  - CHU de Caen-Hopital Cote de Nacre, Caen
  - Hopital Saint Antoine, Créteil
  - Centre Hospitalier de Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Institut Paoli-Calmettes, Marseille
  - Hopital Tenon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Toulouse-Hopital Larrey, Toulouse
  - Institut Gustave Roussy, Villejuif
- South Korea (8):
  - Chungbuk National University Hospital, Cheongju-si
  - The Catholic University of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun Jeonnam
  - National Cancer Center, Korea
  - Seoul National University Bundang Hospital, Seongnam
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Quiron Dexeus Barcelona, Barcelona
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga